CLINICAL TRIAL: NCT00004479
Title: Randomized Study of Midodrine, an Alpha Adrenergic Agonist, in Patients With Neurally Mediated Syncope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14181; MTS-GCO-97-160NE; ROBERTS-MTS-GCO-97-160NE
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Syncope
Keywords: neurologic and psychiatric disorders; rare disease; syncope
MeSH Terms: conditions — Syncope; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Midodrine

INTERVENTIONS:
Drug: midodrine

SUMMARY:
OBJECTIVES:

Determine the efficacy of midodrine, a selective alpha 1 adrenergic agonist, in preventing neurally mediated syncope.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind, crossover, placebo-controlled study.

On day one, patients receive either midodrine or placebo. On day three, patients receive the opposite drug.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Diagnosis of neurally mediated syncope (vasovagal fainting) Sudden fall in blood pressure AND Slowing of the heart AND Temporary loss of consciousness AND Hemodynamic response to head up tilt --Prior/Concurrent Therapy-- No other concurrent adrenergic agonist or antiagonist --Patient Characteristics-- Fertile patients must use effective birth control

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States